CLINICAL TRIAL: NCT00907452
Title: Pharmacogenomic Study to Predict Survival, Best Response and Toxicity in Newly Diagnosed Myeloma Patients Above the Age of 65 Treated With Either a Combination of Melphalan-prednisone-thalidomide or Lenalidomide-dexamethasone
Brief Title: Pharmacogenomic Study in Myeloma Patients Treated With Melphalan-prednisone-thalidomide or Lenalidomide-dexamethasone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intergroupe Francophone du Myelome (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IFM 2007-03; Eudract: 2008-003486-58
Record Dates: First submitted 2009-05-20; First posted 2009-05-22 (Estimated); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Myeloma
Keywords: Pharmacogenomics; prediction response; prediction adverse event
MeSH Terms: conditions — Neoplasms, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- melphalan-prednisone-thalidomide (Active Comparator)
  Interventions: Drug: melphalan-prednisone-thalidomide
- lenalidomide-dexamethasone (Active Comparator)
  Interventions: Drug: lenalidomide-dexamethasone

INTERVENTIONS:
Drug: melphalan-prednisone-thalidomide
  Arms: melphalan-prednisone-thalidomide
Drug: lenalidomide-dexamethasone
  Arms: lenalidomide-dexamethasone

SUMMARY:
This protocol (in patients aged 65 and over suffering from previously untreated multiple myeloma), represents the first worldwide, pharmacogenomic study on this scale in terms of the number of patients analyzed and the implemented molecular diagnostics resources. The goal is to be able to identify patients who will best respond to the study treatments or experience the fewest associated side effects and improve prognosis, in order to optimize care management in multiple myeloma.

To this end, the study seeks to predict the following parameters in these patients:

* The treatment response and occurrence of adverse events linked to a lenalidomide-dexamethasone combination or a melphalan-prednisone-thalidomide combination.
* Progression-free survival and overall survival.

Prediction of the treatment response and the occurrence of adverse effects will be based on:

* An analysis of constitutive genetic traits linked to single nucleotide polymorphisms and DNA copy number variations.
* An analysis of changes in the tumor's genotype (change in the DNA copy number) and phenotype (altered gene and micro-RNA expression).

Prediction of progression-free survival and overall survival will be based on an analysis of changes in the tumor's genotype and phenotype.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form
* Age ≥ 65 years at the time of signing consent
* Previously untreated, symptomatic multiple myeloma as defined by the 3 criteria below: MM diagnostic criteria (all 3 required)

  * Monoclonal plasma cells in the bone marrow ≥10% and/or presence of a biopsy-proven plasmacytoma
  * Monoclonal protein present in the serum and/or urine
  * Myeloma-related organ dysfunction (at least one of the following):

    * Calcium elevation in the blood (serum calcium > 10.5 mg/l or upper limit of normal)
    * Renal insufficiency (serum creatinine > 2 mg/dl)
    * Anemia (hemoglobin < 10 g/dl or 2 g < normal)
    * Lytic bone lesions or osteoporosis
* have measurable disease by protein electrophoresis analyses as defined by the following:

  * IgG multiple myeloma: Serum monoclonal paraprotein (M-protein)level ≥ 1.0 g/dL or urine M-protein level ≥ 200 mg/24 h
  * IgA multiple myeloma: Serum M-protein level ³ 0.5 mg/dL or urine M-protein level³ 200 mg/24 h
  * IgM multiple myeloma (IgM M-protein plus lytic bone disease documented by skeletal survey plain films): Serum M-protein level ≥ 1.0 g/dL or urine Mprotein level ≥ 200 mg/24h
  * IgD multiple myeloma: Serum M-protein level ≥ 0.05 g/dL or urine M-protein level ≥ 200 mg/24h
  * Light chain multiple myeloma: Serum M-protein level ≥ 1.0 g/dL or urine Mprotein level ≥ 200 mg/24 hours
* ECOG performance status of 0, 1, or 2
* Treated by either melphalan-prednisone-thalidomide or lenalidomide- dexamethasone

Exclusion Criteria:

* Previous treatment with antimyeloma therapy (does not include radiotherapy, bisphosphonates, or a single short course of steroid [i.e., less than or equal to the equivalent of dexamethasone 40 mg/day for 4 days; such a short course of steroid treatment must not have been given within 28 days (4 weeks) of randomization]
* Any serious medical condition that places the patient at an unacceptable risk if he or she participates in this study
* Any of the following laboratory abnormalities :

  * Absolute neutrophil count (ANC) < 1,000 cells/µL (1.0 x 109/L)
  * Platelet count < 50,000 cells/µL (50 x 109/L) for patients in whom < 50% of bone marrow nucleated cells are plasma cells; but platelet count < 30,000/µL for patients in whom ≥ 50% of bone marrow nucleated cells are plasma cells
  * Serum SGOT/AST or SGPT/ALT > 3.0 x upper limit of normal (ULN)
  * Creatinine clearance ≤ 30 mL/min (Cockroft-Gault calculation)
* Prior history of malignancies, other than multiple myeloma, unless the subject has been free of the disease for ≥ 3 years. Exceptions include the following:

  * Basal cell carcinoma of the skin
  * Squamous cell carcinoma of the skin
  * Carcinoma in situ of the cervix
  * Carcinoma in situ of the breast
  * Incidental histological finding of prostate cancer (TNM stage of T1a or T1b)
* Patients who have are unable or unwilling to undergo antithrombotic therapy
* Peripheral neuropathy of > grade 2 severity
* Known HIV positivity or active infectious hepatitis, type A, B, or C.
* Primary AL amyloidosis and myeloma complicated by amyloidosis.
* Renal failure requiring dialysis

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 143 (Actual)
Dates: Start 2009-07-29 (Actual); Primary Completion 2010-12-14 (Actual); Study Completion 2016-07-14 (Actual)

PRIMARY OUTCOMES:
best response to treatment | 1 year
  best response rate

CONTACTS AND LOCATIONS:
Overall Officials: Philippe MOREAU, Pr, Study Chair — Departement of clinical Hematology (University Hospital of Nantes)
Locations (26):
- France (26):
  - CH ALBI, Albi
  - CHRU Angers, Angers
  - CH Côte basque, Bayonne
  - CH Blois, Blois
  - BORDEAUX, Bordeaux
  - Chalon sur Saone, Chalon-sur-Saône
  - CHU Dijon, Dijon
  - Ch Dunkerque, Dunkirk
  - Chu Grenoble, Grenoble
  - CHD Vendée, La Roche-sur-Yon
  - CHRU Lille, Lille
  - CHU LYON, Lyon
  - LYON SUD, Lyon
  - Ipc Marseille, Marseille
  - CHR METZ, Metz
  - CH Mulhouse, Mulhouse
  - Chu Nancy, Nancy
  - Chu Nantes, Nantes
  - Centre Antoine LACASSAGNE, Nice
  - Institut Curie, Paris
  - Chu Poitiers, Poitiers
  - Chu Rennes, Rennes
  - CH Yves Le Foll, Saint-Brieuc
  - René Huguenin, Saint-Cloud
  - Chu Toulouse, Toulouse
  - Chu Tours, Tours

REFERENCES:
- [Result] Miannay B, Minvielle S, Roux O, Drouin P, Avet-Loiseau H, Guerin-Charbonnel C, Gouraud W, Attal M, Facon T, Munshi NC, Moreau P, Campion L, Magrangeas F, Guziolowski C. Logic programming reveals alteration of key transcription factors in multiple myeloma. Sci Rep. 2017 Aug 23;7(1):9257. doi: 10.1038/s41598-017-09378-9. PMID 28835615